CLINICAL TRIAL: NCT02858648
Title: Diabetes Go Mobile! - A Pilot Study Testing the Effect of a Behavioral Intervention With Smart Phone Based Self-Monitoring on Glycemic Control and Vascular Inflammatory Markers
Brief Title: Diabetes Go Mobile! Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Harris Health System (Unknown)
Responsible Party: Principal Investigator, Jing Wang, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-SN-12-0582
Record Dates: First submitted 2016-08-02; First posted 2016-08-08 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Behavior intervention with smart phone based self-monitoring (Experimental): Patients in this group were asked to attend 11 group and 1 individual session over 6 months, and received a smartphone with two downloaded applications to monitor diet, physical activity, weight, and blood glucose (connected with a blue tooth glucometer) throughout 6 months.
  Interventions: Behavioral: Behavior intervention with smart phone based self-monitoring
- Behavior intervention with paper diary based self-monitoring (Experimental): Patients in this group were asked to attend 11 group sessions and 1 individual session over 6 months, and received paper diaries along with a calorie counter booklet, weight scale, food scale, and pedometer to monitor diet, physical activity, weight, and blood glucose throughout 6 months.
  Interventions: Behavioral: Behavior intervention with paper diary based self-monitoring
- Usual care (No Intervention): Patients in this group received no intervention, they continue to receive usual diabetes care and education from the recruitment clinic.

INTERVENTIONS:
Behavioral: Behavior intervention with smart phone based self-monitoring — Use two smartphone applications for self-monitoring of diet, physical activity, weight, and blood glucose (connected via a blue-tooth enabled glucometer), plus 11 group session and 1 individual session focused on behavioral strategies
  Arms: Behavior intervention with smart phone based self-monitoring
Behavioral: Behavior intervention with paper diary based self-monitoring — Use paper diaries along with a calorie counter booklet, weight scale, food scale, and pedometer for self-monitoring of diet, physical activity, weight, and blood glucose, plus 11 group session and 1 individual session focused on behavioral strategies
  Arms: Behavior intervention with paper diary based self-monitoring

SUMMARY:
The purpose of this study is to examine whether a behavioral lifestyle intervention using mobile smart phone technology for self-monitoring can lead to greater improvements in diabetes outcomes.

DETAILED DESCRIPTION:
The investigators will conduct a pilot randomized controlled clinical trial to examine the feasibility and preliminary efficacy of a behavioral lifestyle intervention on weight, glycemic control, and vascular inflammatory marker outcomes. A total of 26 overweight or obese patients with type 2 diabetes will be recruited from an underserved minority community health center in Houston, TX. They were randomly assigned into one of the three groups: 1) Behavior intervention with smart phone based self-monitoring, 2) Behavior intervention with paper diary based self-monitoring, and 3) Usual care group. Both Mobile and Paper groups received a total of 11 group sessions and 1 individual session in a 6-month intervention. Mobile group received an android-based smart phone with two applications loaded to help them record their diet, physical activity, weight, and blood glucose, while the paper group is using paper diaries for these recordings.

ELIGIBILITY:
Inclusion Criteria:

* 21 to 74 years of age
* BMI≥ 25 kg/m2
* Self-reported being diagnosed with type 2 diabetes for at least 6 months
* Currently monitor blood glucose and has a blood glucose meter
* Be able to read and write in English

Exclusion Criteria:

* Previously participated in a structured lifestyle intervention, such as Look AHEAD in the last 12 months
* Current pregnant /nursing or plan to become pregnant in the next 6 months
* In addition to their diabetes condition, presence of a current serious illness or unstable condition requiring supervision on a special diet and limiting their ability to perform physical activity level.
* Current treatment for a severe psychological disorder
* Planned vacation, absences, or relocation in the next 6 months

Ages: 21 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in Weight as assessed by the Tanita Scale | baseline, 3 months, 6 months
Change in Glycemic control as assessed by HbA1c levels | baseline, 3 months, 6 months

SECONDARY OUTCOMES:
Change in Dietary intake as measured by the Automated Self-administered 24-hour Dietary Recall (ASA24™) version 1 | baseline, 3 months, 6 months
Change in Physical Activity as assessed by accelerometer | baseline, 3 months, 6 months
Change in Physical Activity as assessed by IPAQ-Short Form | baseline, 3 months, 6 months
Change in Blood pressure as assessed by automated blood pressure cuff | baseline, 3 months, 6 months
Change in Waist circumference | baseline, 3 months, 6 months
Change in Inflammation as assessed by C-reactive protein levels | baseline, 3 months, 6 months
Change in Inflammation as assessed by IL-6 levels | baseline, 3 months, 6 months
Percent attendance at group sessions | 6 months
Percent adherence to self-monitoring | 6 months
Change in Health literacy as measured by the Newest Vital Sign health literacy assessment | baseline, 3 months, 6 months
Change in Medication Adherence as assessed by the Morisky medication adherence questionnaire | baseline, 3 months, 6 months
Change in Depression as measured by the Center for Epidemiologic Studies Depression Scale (CES-D) | baseline, 3 months, 6 months
Change in Diabetes Self-Care as Assessed by the Summary of Diabetes Self-Care Activities Expanded Version | baseline, 3 months, 6 months
Change in Quality of life as assessed by the PROMIS Global | baseline, 3 months, 6 months
Change in Clinical utility as assessed by the PROMIS 57 | baseline, 3 months, 6 months
Change in Perceived Stress as measured by the Perceived Stress Scale | baseline, 3 months, 6 months
Change in Sleep Quality as assessed by the Pittsburgh Sleep Quality Index | baseline, 3 months, 6 months
Change in Sleepiness. Assessed by the Epworth Sleepiness Scale | baseline, 3 months, 6 months
Change in Self-efficacy for diabetes as assessed by the Self-efficacy for diabetes measure | baseline, 3 months, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jing Wang, PhD, MPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jiwani R, Wang J, Berndt A, Ramaswamy P, Mathew Joseph N, Du Y, Ko J, Espinoza S. Changes in Patient-Reported Outcome Measures With a Technology-Supported Behavioral Lifestyle Intervention Among Patients With Type 2 Diabetes: Pilot Randomized Controlled Clinical Trial. JMIR Diabetes. 2020 Jul 24;5(3):e19268. doi: 10.2196/19268. PMID 32706652
- [Derived] Wang J, Cai C, Padhye N, Orlander P, Zare M. A Behavioral Lifestyle Intervention Enhanced With Multiple-Behavior Self-Monitoring Using Mobile and Connected Tools for Underserved Individuals With Type 2 Diabetes and Comorbid Overweight or Obesity: Pilot Comparative Effectiveness Trial. JMIR Mhealth Uhealth. 2018 Apr 10;6(4):e92. doi: 10.2196/mhealth.4478. PMID 29636320